CLINICAL TRIAL: NCT00566423
Title: Biomarkers in the Diagnosis and Assessment of PAH
Brief Title: Biomarkers in the Diagnosis and Assessment of Pulmonary Arterial Hypertension (PAH)
Acronym: Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Arunabh Talwar MD, North Shore-Long Island Jewish Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-030; NS-LIJHS IRB # 07-030
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Biomarkers; MIF; BNP; 6 Minute Walk (6MW)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients with Pulmonary Arterial Hypertension
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Venous and Arterial Blood draw samples; 6 Minute Walk test

SUMMARY:
The investigators hypothesize that baseline plasma brain natriuretic peptide (BNP) and migration inhibitory factor (MIF) levels are surrogate markers of clinical severity of PAH and that changes in plasma brain natriuretic peptide (BNP) and MIF levels pre and post exercise.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PAH, based on currently accepted gold standard for Right Heart Catheterization.
* Patients with mean artery pressure of greater that 25 mm Hg at rest or 30mm Hg during exercise with pulmonary capillary wedge pressure less than 18mm Hg on right heart catheterization.

Exclusion Criteria:

* Significant left heart disease or renal insufficiency (serum creatinine > 1.5 mg%).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assess the correlation of plasma/arterial BNP and MIF levels pre/post with the 6 Minute walk test distance and echocardiographic parameters as surrogate markers of severity of PAH. | 2 year

SECONDARY OUTCOMES:
To determine if changes in plasma/arterial MIF levels pre/post 6MW test are due to MIF released from the lungs | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Arunabh Talwar, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-Long Island Health System, New Hyde Park, New York, United States